CLINICAL TRIAL: NCT05321277
Title: Response of Cardiometabolic Biomarkers and Gut Microbiota to Walnut Consumption
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1867437
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Diseases
Keywords: heart health; gut microbiota; Mediterranean diet; cardiometabolic health; gut health; diet
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walnut diet (Active Comparator): Participants will consume 56 g of walnuts each day at home for 3 weeks.
  Interventions: Dietary Supplement: Walnuts
- No-nut diet (Active Comparator): Participants will follow a no-nut diet for 3 weeks.
  Interventions: Dietary Supplement: No-nut diet

INTERVENTIONS:
Dietary Supplement: Walnuts — Participants will consume 56 g of walnuts daily for 3 weeks. Participants will also follow a diet devoid of ellagitannin-rich, high fiber, and fermented foods.
  Arms: Walnut diet
Dietary Supplement: No-nut diet — Participants will exclude all nuts and nut-derived products; high-fiber, fermented and ellagitannin-rich foods will also be excluded.
  Arms: No-nut diet

SUMMARY:
The purpose of this research is to test if eating walnuts will cause any changes in blood lipids (like good and bad cholesterol, for example) and levels of inflammation in the blood, as well as changes in the bacteria living in the gut.

DETAILED DESCRIPTION:
The purpose of this research is to test if eating walnuts will cause any changes in blood lipids (like good and bad cholesterol, for example) and levels of inflammation in the blood, as well as changes in the bacteria living in the gut. Overweight/obese adults between the ages of 45 and 70 yo with elevated LDL-C levels are eligible to participate. The study involves 5 visits (1 initial screening and 4 study visits) and will last about 10 weeks. There is a 1-week run-in period before starting the study, followed by two diet intervention periods each lasting 3 weeks, separated by a 3-week washout period.

Participation in this study will involve an initial 1-week run in period to become accustomed to the study diet. After this 1 week period, participants will be randomly selected to start either a walnut or a no-nut diet. During each phase of the study, participants will be asked to come to the University of California, Davis campus after a 10-12 hour overnight fast. At each visit, body measurements will be taken; blood, urine and fecal samples will be collected.

During the 10 weeks of the study, all nuts and nut-derived products will need to be avoided. The study will provide walnuts to be eaten at home for each intervention phase. Additionally, the investigators will ask that ellagitannin-rich foods, high-fiber and fermented foods be avoided in the diet. Detailed food diaries will be filled out and brought to study visits.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese men and postmenopausal women between 45-70 years of age, BMI range of 25.0-39.9 kg/m2 and elevated LDL-C levels (130-189 mg/dL).

Exclusion Criteria:

* Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant or lactating women, women planning to become pregnant in the next four months and prisoners will be specifically excluded.

Additional exclusion criteria are listed below:

* Allergy to walnuts or other nuts
* Eating more than 25 grams of fiber per day, assessed by the Block Dietary-Fruit-Vegetable-Fiber Screener©
* Taking medications or supplements known to affect metabolism or gut microbiota composition (i.e. Metformin, statins, antibiotics within the past 3 months, fiber supplements, probiotics, and others)
* Documented chronic diseases including diabetes, renal or liver disease, metabolic syndrome, active cancer, MI or stroke, history of gastric bypass or GI disease (e.g. Crohn's Disease, Irritable Bowel Disease, diverticulosis, diverticulitis, etc.)
* Smoker or living with a smoker, including vaporizer and/or electronic cigarettes.
* Illicit drug use, cannabis usage, or consuming >1 alcoholic drink/day
* Extreme dietary or exercise patterns
* Recent weight fluctuations (>10% in the last 6 months)
* Taking prescription lipid medications or supplements that may affect lipoprotein metabolism (i.e. >1 g of fish oil/day, antioxidant supplements)
* Taking exogenous hormones
* Poor venous access
* Unwillingness to comply with study protocols

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assessing the influence of walnut consumption on blood lipid measurements. | Through study completion, an average of 10 weeks
  Measure for changes in the levels of HDL and LDL in separated plasma; measured in units of mg/dL. Blood will be assessed for the fasting (baseline) sample at each of the 4 study visits.
Assessing the influence of walnut consumption on circulating inflammatory markers: PAI-1, VCAM-1 and ICAM-1. | Through study completion, an average of 10 weeks
  Measure circulating inflammatory markers in separated plasma at each of the 4 study visits. Commercially available ELISA kits will be used: PAI-1, VCAM-1, ICAM-1.
Assessing the influence of walnut consumption on blood pressure. | Through study completion, an average of 10 weeks
  Measure blood pressure (mmHg) before the start of drawing blood on study day protocols.

SECONDARY OUTCOMES:
Assessing the influence of walnut consumption on fecal pH. | Through study completion, an average of 10 weeks
  Measure fecal pH via pH meter at each of the 4 study visits.
Assessing the influence of walnut consumption on stool consistency. | Through study completion, an average of 10 weeks
  Assess fecal consistency using Bristol Stool Scale at each of the 4 study visits. The scale runs from Type 1 (the lowest) to Type 7 (the highest). The desirable Type is either 3 or 4. Types 1 and 2 may be indicative of constipation, while Types 5, 6, and 7 may indicative diarrhea.
Assessing the influence of walnut consumption on fecal moisture. | Through study completion, an average of 10 weeks
  Measure fecal moisture by weighing wt and vacuum dried feces in grams at each of the 4 study visits.
Assessing the influence of walnut consumption on the levels of gut inflammatory markers: Lipocalin-2 and calprotectin. | Through study completion, an average of 10 weeks
  Measure fecal levels of Lipocalin-2 and calprotectin at each of the 4 study visits. Commercially available ELISA kits will be used: lipocalin-2, calprotectin.
Assessing the influence of walnut consumption on plasma and urine levels of walnut-derived metabolites - urolithins. | Through study completion, an average of 10 weeks
  Measure urolithin levels in separated plasma and urine via metabolomics analysis at each of the 4 study visits.

OTHER OUTCOMES:
Food record analysis | Through study completion, an average of 10 weeks
  Use a computer program to check for study dietary requirements. Subjects are to avoid olives and olive containing products during study protocol periods. This will be done using a subject self-recorded 3-day food record submitted to study personnel.
Anthropometric measurements | Through study completion, an average of 10 weeks
  Measure waist (cm) and hip circumference (cm) before the start of drawing blood on study day protocols.
Measure of changes in weight | Through study completion, an average of 10 weeks
  Measure weight (kg) before the start of drawing blood on study day protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Ragle Human Nutrition Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No